CLINICAL TRIAL: NCT06645353
Title: Evaluation of Perfusion and Oxygenation in Muscle of Patients With PAD Undergoing LER
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: iThera Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MSOT
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MSOT Multispectral Optoacoustic Tomography — MSOT Multispectral Optoacoustic Tomography, single-wavelength, HbT, Hb, HbO2, collagen and mSO2 (700-1.100 nm wavelength range, in 10 nm increments) in the tibialis anterior and flexor hallucis brevis, at multiple time-points before, during and after interventional LER Lower Extremity Revascularization .

SUMMARY:
During this IIT, the MSOT (Multispectral Optoacoustic Tomography ) Acuity Echo will be used to scan participants with Peripheral Arterial Disease assess MSOT Multispectral Optoacoustic Tomography (single-wavelength and hemoglobin-related parameters) in the Tibialis Anterior, and flexor hallucis brevis, at multiple time-points before, during and after interventional Lower Extremity Revascularization (LER ).

Primary aim of the study ist the Comparison of the difference between oxygenated, deoxygenated hemoglobin and oxygenation in the tibialis anterior, and flexor hallucis brevis, at multiple time-points before, during and after interventional Lower Extremity Revascularization.

ELIGIBILITY:
Inclusion Criteria:

* • Written consent of the participant after being informed

  * Adults above 18 years
  * Participants with PAD stage 4 - 6 (Rutherford) with indication for interventional LER

Exclusion Criteria:

* • Participants with previous LER on the same leg

  * Participants less than 18years
  * Pregnancy
  * Participants with tattoos in the scan area
  * Participants with no clinical indication for interventional LER
  * Missing consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • Participants with PAD stage 4 - 6 (Rutherford) with indication for interventional LER
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
MSOT Multispectral Optoacoustic Tomography, | baseline pre LER, 30 minutes post LER, 24 hours post LER, 48hours post LER
  single-wavelength, HbT, Hb, HbO2, collagen and mSO2 (700-1.100 nm wavelength range, in 10 nm increments) in the tibialis anterior and flexor hallucis brevis, at multiple time-points before, during and after interventional LER Lower Extremity Revascularization .

IPD SHARING:
Plan to Share IPD: No